CLINICAL TRIAL: NCT00606177
Title: A Multicenter, Placebo-controlled, Double-blind Investigative Extension Trial of the Safety and Efficacy of Aripiprazole in the Treatment of Patients With Bipolar Disorder Experiencing a Manic or Mixed Episode
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-06-004
Record Dates: First submitted 2008-01-19; First posted 2008-02-01 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-01

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Aripiprazole
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aripiprazole — oral, 24mg(4 tablets)/day
  Other Names: OPC-14597
  Arms: 1
Drug: placebo — oral, 0mg(4tablets)/day
  Other Names: OPC-14597
  Arms: 2

SUMMARY:
To investigate the safety and efficacy of long-term administration of aripiprazole by performing extended administration of the treatment administered in the preceding multicenter, double-blind, placebo-controlled, parallel group-comparison trial of aripiprazole in patients with bipolar disorder experiencing a manic or mixed episode (Study 031-06-003, hereafter "Study 003") in a double-blind manner to those patients who complete Study 003 and demonstrate drug efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Trial subjects will be men and women of age 18 or above and below the age of 65 who will not be turning 65 during the trial.
* Subjects have the ability to understand and to provide informed consent to the examination, observation, and evaluation processes specified in this protocol, and have signed the informed consent form based on a full understanding of the trial.
* Subjects who meet DSM-IV-TR criteria for manic or mixed episodes and have been diagnosed as having "296.4x Bipolar I Disorder in which the most recent episode was manic" or "296.6x Bipolar I Disorder in which the most recent episode was mixed"
* Subjects who were enrolled in and have completed Study 003 and who meet the following criteria for demonstration of drug efficacy
* Subjects demonstrating drug efficacy:

  * Those subjects who completed Study 003 whose score for CGI-BP Change From Preceding Phase (mania) at the time of evaluation on Day 21 of Study 003 (completion) was between 1 (Very much improved) and 3 (Minimally improved)

Exclusion Criteria:

* Subjects presenting with a clinical picture and/or history that is consistent with a DSM-IV-TR diagnosis of:

  * Delirium, dementia, amnestic disorder, or other cognitive disorders
  * Schizophrenia or other psychotic disorder
  * Personality disorder
* Subjects with psychotic symptoms that are clearly due to another general medical condition or direct physiological effects of a substance
* Subjects who represent a significant risk of committing suicide
* Subjects known to have a complication of allergy to aripiprazole or other quinolinone-skeleton compounds
* Subjects with a complication of neuroleptic malignant syndrome
* Subjects in a state of physical exhaustion accompanied by such conditions as dehydration or malnutrition
* Subjects with a complication of paralytic ileus
* Subjects with a complication of organic brain disorder or convulsive disorder, such as epilepsy
* Subjects with a complication of diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Department of Clinical Research and Development, Division of New Product Evaluation and Development
Locations (12):
- Hong Kong, China
- Japan (9):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Hokuriku Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region
- Seoul, South Korea
- Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: Patients who had completed the preceding study and demonstrated drug efficacy were the target.
  Subjects were administered 24 ,12, or 30 mg/day of aripiprazole once daily for 154 days.
- Placebo: Patients who had completed the preceding study and demonstrated drug efficacy were the target.
  Subjects were administered placebo once daily for 154 days.
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 55 | 44
Completed | 28 | 19
Not Completed | 27 | 25
Not completed — Adverse Event | 9 | 5
Not completed — Lack of Efficacy | 3 | 7
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 4
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Progression to depressive phase | 6 | 1
Not completed — Diabetic blood glucose level/ High HbA1c | 1 | 1
Not completed — Change of residence or other commitments | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Population(FAS)：Excluding 3 subject with GCP violation from the randomized subjects.
  (Aripiprazole:1, Placebo:2)
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 54 | 42 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (11.95) | 37.8 (11.67) | 38.3 (11.78)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 54 | 41 | 95
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 53
  Male | 25 | 18 | 43
Region of Enrollment [Number; unit: participants]
  Taiwan | 4 | 9 | 13
  China | 9 | 9 | 18
  Japan | 22 | 10 | 32
  Malaysia | 4 | 6 | 10
  Indonesia | 5 | 2 | 7
  Philippines | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: Using LOCF datasets, descriptive statistics of actual values for changes of YMRS total scores from baseline (Day 1 of preceding study) to endpoint (Day 154) was calculated for each treatment group.
  YMRS is composed of 11 evaluation items with 5 rating levels each. Items rated on a scale of 0 to 4 (comprising 5 rating levels of one point each) are 1) levated mood, 2) increased motor activity/energy, 3) sexual interest, 4) sleep, 7) language-thought disorder, 10) appearance, and 11) insight. Items rated on a scale of 0 to 8 (comprising 5 rating levels of two points each) are 5) irritability, 6) speech (rate and amount), 8) content, and 9) disruptive-aggressive behavior.
  YMRS ranges from 0 (best possible outcome) to 60 (worst possible outcome).
Time Frame: Baseline (Day 1 of preceding study) , Day 154 or at discontinuation
Population: FAS: The FAS consisted of subjects who had received at least one dose of investigational product and for whom the post-dosing efficacy parameter data had been obtained. Cases of GCP violation were excluded from analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 54 | 42
scores on a scale | -22.6 (11.08) | -15.4 (12.90)

2. Secondary Outcome: Clinical Global Impression - Bipolar Version (CGI-BP) Severity of Illness (Mania)
Description: Using LOCF datasets, descriptive statistics of actual values for change of CGI-BP severity of illness score (mania) from baseline (Day 1 of preceding study) to endpoint (Day 154) were calculated for each treatment group.
  CGI-BP severity of illness is a scale for overall evaluation of the severity of bipolar disorder; it comprises 3 components-mania, depression, and overall bipolar illness.
  CGI-BP severity of illness score (mania) ranges form 1 (normal, not ill) to 7 (very severely ill).
Time Frame: Baseline (Day 1 of preceding study), Day 154 or at discontinuation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 54 | 42
scores on scale | -2.9 (1.45) | -1.9 (1.70)

ADVERSE EVENTS:
Time Frame: 22 weeks
Arm/Group | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 7/54 | 4/42
Other Adverse Events (participants affected / at risk) | 46/54 | 26/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=54) | Placebo (N=42)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Stupor (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Bipolar I Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 1 (1)
Bipolar Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delusion of Grandeur (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=54) | Placebo (N=42)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 4 (6)
Salivary Hypersecretion (Gastrointestinal disorders) | 6 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 6 (11)
Toothache (Gastrointestinal disorders) | 3 (5) | 2 (3)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 5 (6) | 5 (6)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (4) | 5 (5)
Excoriation (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Weight Increased (Investigations) | 9 (9) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 3 (3) | 0 (0)
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Akathisia (Nervous system disorders) | 17 (20) | 7 (8)
Tremor (Nervous system disorders) | 10 (11) | 4 (7)
Headache (Nervous system disorders) | 2 (2) | 5 (6)
Dizziness (Nervous system disorders) | 2 (2) | 4 (6)
Bradykinesia (Nervous system disorders) | 5 (6) | 0 (0)
Dyskinesia (Nervous system disorders) | 3 (4) | 1 (1)
Somnolence (Nervous system disorders) | 3 (4) | 1 (2)
Insomnia (Psychiatric disorders) | 7 (7) | 7 (13)
Mania (Psychiatric disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No